CLINICAL TRIAL: NCT07231575
Title: Preoperative Stereotactic Body Radiotherapy and Tislelizumab (Immunotherapy) Plus Anlotinib for Operable Stage IB to III EGFR Wild-type Non-small Cell Lung Cancer（STATION）
Brief Title: Neoadjuvant SBRT and Tislelizumab (Immunotherapy) Plus Anlotinib for Resectable EGFR Wild-type NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianhua Fu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STATION
Record Dates: First submitted 2025-07-05; First posted 2025-11-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Neoadjuvant Immunotherapy; NSCLC; Chemo-free Therapy
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Stereotactic body radiotherapy and Tislelizumab (immunotherapy) plus Anlotinib (Experimental)
  Interventions: Radiation: SBRT; Drug: Immunotherapy; Drug: antiangiogenesis therapy

INTERVENTIONS:
Radiation: SBRT — SBRT 8Gy*3
Drug: Immunotherapy — Tislelizumab (immunotherapy) 200mg Q3W
Drug: antiangiogenesis therapy — Anlotinib 8mg D1-D14 Q3W

SUMMARY:
The neoadjuvant strategy of immunotherapy combined with chemotherapy has been recommended for resectable or potentially resectable tumors without driver-gene alterations.However, the AE of chemotherapy is more than 40%，which bring fear to the patients，especially for those who cannot tolerate or refuse chemotherapy.Several studies indicated that the strategies of chemo-free ,such as the combination of immunotherapy with antiangiogenic therapy or with SBRT, were safe and well tolerated, without increasing adverse reactions. Both of them have a promising efficacy with a manageable toxicity profile in patients with resectable NSCLC. The investigators aim to assess the activity and safety of neoadjuvant SBRT and immunotherapy plus antiangiogenic therapy in patients with resectable NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1.18 years or older 2. Eastern Cooperative Oncology Group performance status: 0 or 1 3. Clinical stage IB to IIIB (T3-4N2) Resectable NSCLC 4. Adequate cardiopulmonary and haematological function.

Exclusion Criteria:

1. Known EGFR-sensitising mutations and EML4-ALK fusions
2. Concomitant malignancy, history of another cancer within the past 3 years.
3. Current or previous use of immunosuppressive medication,active autoimmune disease, and interstitial lung disease or idiopathic pulmonary fibrosis on a screening radiographic scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2032-05-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response(pCR, rate) | At the time of surgery

SECONDARY OUTCOMES:
Major pathologic response rate(MPR rate)，Disease-free survival（DFS, month），Event-free survival（EFS,month） | Major Pathologic Response (MPR, rate ):At the time of surgery Disease-Free Survival（DFS, month):From enrollment to disease recurrence or death from any cause Event-Free Survival（EFS,month）：From enrollment to the first pre-specified event

IPD SHARING:
Plan to Share IPD: No